CLINICAL TRIAL: NCT04292028
Title: The Effects of Clinical Pilates Training on Disease-specific Indices, Core Stability, and Balance in Patients With Ankylosing Spondylitis
Brief Title: The Effects of Clinical Pilates Training in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Yasemin ACAR, Research assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/07-33
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; pilates; postural balance; physical endurance; flexibility
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates group (Experimental): The Pilates group participated in an 8-week clinical Pilates training program
  Interventions: Other: Pilates
- Control group (Active Comparator): Control group were given a home-based exercise program
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Pilates — The Pilates group participated in an 8-week clinical Pilates training program
  Arms: pilates group
Other: Home exercises — Control group were given a home-based exercise program.
  Arms: Control group

SUMMARY:
The objective of this study was to examine the effects of 8-week clinical Pilates training on disease-specific indices, core stability, and balance in ankylosing spondylitis (AS) patients.

DETAILED DESCRIPTION:
The objective of this study was to examine the effects of 8-week clinical Pilates training on disease-specific indices, core stability, and balance in ankylosing spondylitis (AS) patients. AS patients were randomly assigned to either the Pilates group (PG) or control group (CG). The PG participated in Pilates training 3 times a week for 8 weeks. Patients in the CG were instructed to follow a home exercise program 3 times a week for 8 weeks. Assessments were performed before and after the interventions. Outcome measures were disease-specific indices, core endurance, and balance. Disease-specific indices were: Bath AS Disease Activity Index (BASDAI), Bath AS Functional Index (BASFI), Bath AS Spinal Mobility Index (BASMI), and the AS Quality of Life (ASqOL) questionnaire. Static core endurance was assessed with trunk flexor, extensor endurance, and lateral side bridge tests, while dynamic core endurance was assessed using modified sit-up test. Balance was assessed with static, dynamic, and single-leg stance postural stability (PS) and limits of stability (LOS) tests using the Biodex Balance System SD.

ELIGIBILITY:
Inclusion Criteria:

* having AS diagnosis based on modified New York criteria,
* being 20-60 years of age, volunteering to participate in the study,
* having no regular exercise habit in the last 6 months,
* agreeing not to participate in any other type of physical exercise program during the study

Exclusion Criteria:

* not attending 4 consecutive Pilates or home exercise sessions,
* change in medication within the previous 6 months or during the study,
* presence of neurological or coexistent systemic disease, history of orthopedic surgery, and active enthesitis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Sponsylitis Disease Activity Index (BASDAI) | 2 minutes
  Disease activity was assessed with the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The index includes patient-reported levels of back pain, fatigue, peripheral joint pain and swelling, localized tenderness, and the duration and severity of morning stiffness. It gives a score ranging from 0-10. High score indicates an increase in disease activity.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 4 minutes
  Functional status was assessed with BASFI. BASFI is comprised of ten items, eight questioning the activities of daily living and two the patient's ability to cope with everyday life. Each is answered on a 10-cm horizontal visual analogue scale (VAS). Total score ranges between 0 and 10, higher scores indicating more severe impairment.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 7 minutes
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) was used to assess spinal mobility. BASMI consists of clinical measures of cervical rotation, tragus wall distance, lumbal flexion (modified Schober) and intermalleolar distance.
Ankylosing Spondylitis Quality of Life (ASQoL) | 3 minutes
  Quality of life was assessed with the Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire, which is the most frequently used disease-specific measure of health-related quality of life. High scores in this 18-item questionnaire indicate severe impairment in quality of life.

SECONDARY OUTCOMES:
Trunk flexor endurance test | 5 minutes
  For trunk flexor endurance test, participants lean on a support which kept the trunk at 60° flexion. Both the knees and hips were flexed to 90°, arms crossed over the chest with the hands placed on the opposite shoulder and feet were fixed. The support of the trunk was then removed, and the participant remained in this position for as long as possible. The test ended when the participant was no longer able to hold the position. The position holding time was recorded in seconds.
Trunk extensor endurance test | 5 minutes
  The extensor endurance test was conducted when the participant lay on the examining table in the prone position with the upper edge of the iliac crests aligned with the edge of the table. The lower body was fixed to the table by two straps, located around the knees and ankles. With the arms folded across the chest, the participant was asked to maintain the upper body in a horizontal position. The time during which the participant could hold this position was recorded in seconds
Side bridge test | 5 minutes
  The lateral side bridge test was performed in the sidelying position on the mat. The subject's knees were extended with the top foot placed in front of the lower foot. The subject supported their weight only on their lower elbow and feet while lifting their hips off the mat. Upper arm crossed over the chest with hand placed on the opposite shoulder. The test ended when the side-lying position was lost, and the position-holding time was recorded in seconds.
Sit-up test | 2 minutes
  Sit-up test was used to assess dynamic core endurance.The subject was positioned supine with knees flexed and feet secured. The arms were crossed on the chest with the hands on the opposite shoulders. To complete a full sit-up, the participant's scapulae touched the mat in the lying position, and the elbows touched the thighs while sitting. The number of correctly executed sit-ups within 60 s was recorded.
Balance Assessment | 10 minutes
  Balance was assessed using the Biodex Balance System SD (Biodex, Inc, Shirley, NY), an instrument designed to measure and train postural stability on a static or unstable surface. . Static postural stability (Level 12, stable platform), dynamic postural stability (Level 4, unstable platform), single-leg stance postural stability (Level 12, stable platform), and limits of stability (LOS) (Level 12, stable platform) tests were performed.

CONTACTS AND LOCATIONS:
Overall Officials: NURSEN İLÇİN, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Acar Y, Ilcin N, Gurpinar B, Can G. The effects of clinical pilates training on disease-specific indices, core stability, and balance in patients with ankylosing spondylitis. J Bodyw Mov Ther. 2023 Jan;33:69-75. doi: 10.1016/j.jbmt.2022.09.010. Epub 2022 Sep 23. PMID 36775528